CLINICAL TRIAL: NCT01371955
Title: Impact of c242T Polymorphism of p22phox in the Development of Diabetic Nephropathy,in Caucasian Diabetic Type 1 Patient.
Brief Title: Impact of c242T Polymorphism of p22phox in Diabetic type1 Nephropathy
Acronym: NEPHRODIANOX
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 1020; 2010-A01074-35 (Registry Identifier: ID RCB)
Record Dates: First submitted 2011-06-10; First posted 2011-06-13 (Estimated); Last update posted 2013-11-15 (Estimated); Status verified 2013-11

CONDITIONS: Type 1 Diabetes Mellitus; Diabetic Nephropathy
Keywords: diabetic nephropathy; CYBA; p22phox; RAGE; 12LOX; genetic; Type 1 Diabetes Mellitus with Diabetic Dermatitis; caucasian; more than twenty years of diabetes duration; older than 18 years; no nephropathy other than diabetic nephropathy
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetic Nephropathies; Granulomatous Disease, Chronic, Autosomal Recessive, Cytochrome B-Negative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We will include 60 patients to reach the required number. We take 2 blood samples: one for genetic analysis and one to determine HBA1c and plasma creatinine. We also take one urinary sample to determine the urinary albumine / creatinine ratio
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- diabetic nephropathy group: patient with diabetic nephropathy, defined as Albuminuria > 30 mg/day or urinary Albumine/ creatinine ratio > 3 mg/mmol ; or GFR estimated by MDRD less than 60 ml/min.1,73m². With no other etiology of diabetic nephropathy.
- diabetic retinopathy group: patient with diabetic retinopathy defined as showing at least one micro aneurysm on retinography. Without nephropathy defined as above
- no complication group: patient without diabetic nephropathy or retinopathy

SUMMARY:
The physiopathology of diabetic nephropathy (DN) is unclear. To investigate risk factor, the investigators choose to look about some oxidative stress genes. Today a one-gene explanation is not really possible. So the theory of some genetic predisposition to DN is more likely.

The aim of the study is to look about the association of the C282T polymorphism of P22phox, a sub unit of the nicotinamide adenine dinucleotide phosphate-oxidase (NADPH oxidase) in the occurrence of DN. To follow the oxidative stress pathway of the DN, the investigators also investigate three other polymorphisms: -429 T/C, -374 T/A polymorphism of advanced glycation end-products receptor (AGER) and the p.Arg261Gln polymorphism of the 12 lipoxygenase (ALOX 12). Discordant data suggest a link between the first 2 polymorphisms and DN. The last polymorphism is correlated to albuminuria in diabetic patients.

DETAILED DESCRIPTION:
To avoid confounding factors, we choose type 1 diabetic patients. We plan, with the data of literature a number need to be significative with a power of 80% and an Alpha risk at 5%, the inclusion of 160 patients for our primary analyze of p 22 phox. Those patients are included consequentially from the diabetic consultation of the university hospital of Grenoble, if they have a history of more than 20 years of diabetes. Those patients have been separated according to the existence of DN, and their polymorphism. Then we estimate with the Fisher test the prevalence of DN in risky patient, and the prevalence of the risky phenotype in the nephropathic patients. Then we investigate with the same statistical test the -429 T/C,he -374 T/A AGER and p.Arg261Gln 12 ALOX polymorphisms.

ELIGIBILITY:
Inclusion Criteria:

* caucasian
* diabetic type 1
* older than 18 years old
* written consent

Exclusion Criteria:

* other etiology of diabetic nephropathy
* pregnancy
* other type of diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: caucasian diabetic type 1 patients with more than 20 years of diabetes duration
Sampling Method: Probability Sample
Enrollment: 162 (Actual)
Dates: Start 2011-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
comparison of prevalence of homozygous polymorphism between the DN-group and the non-DN group | on day 1

SECONDARY OUTCOMES:
comparison of polymorphism of p22phox between the ND group and the sub-group of non-ND patients with diabetic retinopathy only | day 1
comparison of polymorphism prevalence between the 3 groups | day 1
delay between diabetes diagnosis and ND onset by genetic polymorphism | 20 years
  Kaplan Meier method

OTHER OUTCOMES:
albuminuria | day 1
  mg/day
HbA1c | day 1
  HbA1c in %

CONTACTS AND LOCATIONS:
Overall Officials: BENHAMOU pierre yves, MD PhD, Principal Investigator — service de diabétologie
Locations (1):
- University Hospital of Grenoble, Grenoble, France